CLINICAL TRIAL: NCT03852472
Title: A Randomized , Double-Blind, Placebo-Controlled, Parallel Group, Phase 2 Study to Evaluate the Safety and Efficacy of Avacopan in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Evaluation of Safety and Efficacy of Avacopan in Subjects With Moderate to Severe Hidradenitis Suppurativa (AURORA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL016_168
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa
Keywords: Avacopan; ChemoCentryx; Skin Disease; Inflammatory nodule; Abscess; Sinus formation; Fistula formation
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases; Abscess | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Placebo Comparator): Placebo twice daily (BID) for Period 1 of the study
  Interventions: Other: Placebo
- Group B (Experimental): Avacopan 10 mg twice daily (BID) for Period 1+2 of the study
  Interventions: Drug: Avacopan
- Group C (Experimental): Avacopan 30 mg twice daily (BID) for Period 1+2 of the study
  Interventions: Drug: Avacopan
- Placebo to Avacopan 10 mg (Experimental): Treatment period 2, subjects randomized to placebo during period 1 were rerandomized 1:1 to receive 10 mg or 30 mg avacopan BID in period 2.
  Interventions: Drug: Avacopan
- Placebo to Avacopan 30 mg (Experimental): Treatment period 2, subjects randomized to placebo during period 1 were rerandomized 1:1 to receive 10 mg or 30 mg avacopan BID in period 2.
  Interventions: Drug: Avacopan

INTERVENTIONS:
Drug: Avacopan — Active treatment
  Other Names: CCX168
  Arms: Group B; Group C; Placebo to Avacopan 10 mg; Placebo to Avacopan 30 mg
Other: Placebo — Placebo
  Arms: Group A

SUMMARY:
Phase 2 study of Avacopan in Subjects with Moderate to Severe Hidradenitis Suppurativa

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 2 study in subjects with moderate to severe Hidradenitis Suppurativa.

The study is multicenter and will consist of three subject groups. Subjects will be randomized 1:1:1 to a treatment of 10mg avacopan twice daily, 30 mg avacopan twice daily or placebo twice daily for 12 weeks.

Following the 12 weeks double-blind treatment period, subjects on placebo will be re-randomized 1:1 to receive 10 mg or 30 mg avacopan twice daily for additional 24 weeks. Subjects treated with avacopan will continue to receive the same dose (either 10 mg or 30 mg twice daily) for additional 24 weeks.

Subjects will be on study treatment for 36 weeks and will be followed for 44 weeks for assessment of safety and efficacy.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

Primary efficacy analysis will be at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Clinical diagnosis of HS (Hurley Stage II or III), confirmed by a dermatologist, for at least 6 months prior to Screening
* HS lesions are present in at least 2 distinct anatomic areas
* Inadequate or loss of response to a systemic course of antibiotics typically of at least 90 days
* Must have at least 5 inflammatory nodules or abscesses at screening
* Use adequate birth control for subject and partners of child bearing potential
* Willing and able to give written Informed Consent

Exclusion Criteria:

* Pregnant or breast-feeding
* Any other skin disease that may interfere with the assessment of HS
* Rapidly progressive, expanding HS within 30 days prior to screening
* More than 20 draining fistulae at screening
* Any anti-TNF-α treatment for HS or for other conditions prior to Day 1 visit will be prohibited. Exception: Subjects who were previously treated with an anti-TNF-α drug and discontinued treatment >12 weeks prior to Day 1 visit are allowed for enrollment
* Systemic antibiotics are generally excluded
* Topical antibiotics use within 14 days prior to Day 1 is excluded
* Have started a topical prescription medicine for HS within 14 days prior to screening
* A systemic medicine for HS, including biologics and other systemic therapies
* Have received within 14 days prior to Day 1 visit or is expected to require oral or transdermal opioid analgesics (except for tramadol) for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (78):
- United States (78):
  - Clinical Site, Birmingham, Alabama
  - Clinical Site, Mobile, Alabama
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Scottsdale, Arizona
  - Clinical Site, Fort Smith, Arkansas
  - Clinical Site, Rogers, Arkansas
  - Clinical Site, Fountain Valley, California
  - Clinical Site, Fremont, California
  - Clinical Site, Fullerton, California
  - Clinical Site, Huntington Beach, California
  - Clinical Site, Inglewood, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, Manhattan Beach, California
  - Clinical Site, Newport Beach, California
  - Clinical Site, Northridge, California
  - Clinical Site, Redwood City, California
  - Clinical Site, Thousand Oaks, California
  - Clinical Site, Walnut Creek, California
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Clearwater, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Hollywood, Florida
  - Clinical Site, Homestead, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Ocala, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Pembroke Pines, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Weston, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Marietta, Georgia
  - Clinical Site, Newnan, Georgia
  - Clinical Site, Sandy Springs, Georgia
  - Clinical Site, Boise, Idaho
  - Clinical Site, Skokie, Illinois
  - Clinical Site, Crown Point, Indiana
  - Clinical Site, Evansville, Indiana
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Louisville, Kentucky
  - Clinical Site, Metairie, Louisiana
  - Clinical Site, New Orleans, Louisiana
  - Clinical Site, Largo, Maryland
  - Clinical Site, Beverly, Massachusetts
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Quincy, Massachusetts
  - Clinical Site, Clarkston, Michigan
  - Clinical Site, Fort Gratiot, Michigan
  - Clinical Site, Saint Joseph, Michigan
  - Clinical Site, Troy, Michigan
  - Clinical Site, Minneapolis, Minnesota
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Omaha, Nebraska
  - Clinical Site, Verona, New Jersey
  - Clinical Site, New York, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Chapel Hill, North Carolina
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Wilmington, North Carolina
  - Clinical Site, Athens, Ohio
  - Clinical Site, Bexley, Ohio
  - Clinical Site, Cleveland, Ohio
  - Clinical Site, Marion, Ohio
  - Clinical Site, Mason, Ohio
  - Clinical Site, Norman, Oklahoma
  - Clinical Site, Portland, Oregon
  - Clinical Site, Drexel Hill, Pennsylvania
  - Clinical Site, Hershey, Pennsylvania
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Warwick, Rhode Island
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Nashville, Tennessee
  - Clinical Site, Austin, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Sugar Land, Texas
  - Clinical Site, Spokane, Washington
  - Clinical Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Period 1- Placebo BID for 12 Weeks
Period: Period 1 - 12 Weeks
Arm/Group | Group A | Group B | Group C | Placebo to Avacopan 10 mg | Placebo to Avacopan 30 mg
Started (The Intent-to-Treat Population in period 1 (ITT1) was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1 and excluded Site 138 subjects (please see additional milestone below for exact figures)) | 130 | 134 | 134 | 0 (Arm is an extension of Group A from Period 1) | 0 (Arm is an extension of Group A from Period 1)
Excluded Site 138 Subjects From ITT1 (Subjects from Site 138 were excluded from the analysis due to potential misconduct and noncompliance at this site.) | 13 | 11 | 13 | 0 | 0
Completed | 109 | 108 | 109 | 0 | 0
Not Completed | 21 | 26 | 25 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 10 | 7 | 0 | 0
Not completed — Subject noncompliance with dosing or diary completion | 0 | 1 | 3 | 0 | 0
Not completed — Lost to Follow-up | 5 | 5 | 7 | 0 | 0
Not completed — Noncompliance with the protocol | 2 | 0 | 4 | 0 | 0
Not completed — At the discretion of the investigator or sponsor for any reason | 0 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 6 | 4 | 0 | 0
Not completed — Reason not stated | 2 | 1 | 0 | 0 | 0
Period: Period 2 - Week 44
Arm/Group | Group A | Group B | Group C | Placebo to Avacopan 10 mg | Placebo to Avacopan 30 mg
Started (The Intent-to-Treat Population in period 2 (ITT2) was defined as all subjects who received at least 1 dose of investigational product during period 2 and excluded Site 138 subjects (please see additional milestone below for exact figures)) | 0 (In Period 2 this arm becomes Placebo to Avacopan 10mg and Placebo to Avacopan 30mg arms.) | 108 | 108 (As per ITT2 population, 108 participants were enrolled from period 1.) | 56 (As per ITT2 population, 56 participants were enrolled from period 1, previous Group A.) | 53 (As per ITT2 population, 53 participants were enrolled from period 1, previous Group A.)
Excluded Site 138 Subjects From ITT2 (Subjects from Site 138 were excluded from the analysis due to potential misconduct and noncompliance at this site.) | 0 | 7 | 9 | 3 | 6
Completed Week 36 | 0 | 71 | 79 | 41 | 36
Completed Week 44 | 0 | 70 | 75 | 39 | 35
Completed | 0 | 70 | 75 | 39 | 35
Not Completed | 0 | 38 | 33 | 17 | 18
Not completed — Withdrawal by Subject | 0 | 22 | 15 | 10 | 10
Not completed — Subject noncompliance with dosing or diary completion | 0 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 8 | 12 | 1 | 2
Not completed — Noncompliance with the protocol | 0 | 2 | 1 | 0 | 0
Not completed — At the discretion of the investigator or sponsor for any reason | 0 | 1 | 3 | 2 | 3
Not completed — Adverse Event | 0 | 3 | 1 | 2 | 2
Not completed — COVID-19 Related | 0 | 0 | 0 | 1 | 0
Not completed — Reason not stated | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 130 | 134 | 134 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (11.87) | 36.0 (12.05) | 36.8 (11.57) | 36.6 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 28 | 81
  Male | 107 | 104 | 106 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 22 | 39 | 92
  Not Hispanic or Latino | 99 | 112 | 95 | 306
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 43 | 46 | 34 | 123
  White | 83 | 82 | 96 | 261
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 3 | 3 | 2 | 8
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline characteristic value is not available for all patients.
  cm
    number analyzed (Participants) | 129 | 134 | 134 | 397
    (all) | 166.69 (8.696) | 168.67 (9.852) | 167.66 (9.021) | 167.69 (9.221)
Weight [Mean (Standard Deviation); unit: kg] | 102.48 (23.425) | 103.02 (27.817) | 103.46 (28.601) | 102.99 (26.678)
BMI [Mean (Standard Deviation); unit: kg/m²] — BMI - body mass index Population: Baseline characteristic value is not available for all patients.
  kg/m²
    number analyzed (Participants) | 129 | 134 | 134 | 397
    (all) | 36.87 (8.824) | 36.14 (8.728) | 36.75 (9.384) | 36.58 (8.969)
Hurley Stage of HS [Count of Participants; unit: Participants] — HS- Hidradenitis Suppurativa Hurley stage; higher stage indicates more serious disease
  Participants
    Stage II | 85 | 84 | 87 | 256
    Stage III | 45 | 50 | 47 | 142
HS Disease Duration from Time of Diagnosis [Mean (Standard Deviation); unit: years] — HS- Hidradenitis Suppurativa
  years | 11.06 (10.275) | 10.64 (8.733) | 11.21 (9.521) | 10.97 (9.502)
Number of AN Count [Mean (Standard Deviation); unit: abscess and inflammatory nodules] — AN- abscess and inflammatory nodule
  abscess and inflammatory nodules | 11.6 (9.83) | 13.5 (13.41) | 12.3 (9.62) | 12.5 (11.10)
Number of Draining Fistulae [Mean (Standard Deviation); unit: Draining Fistulae] | 2.8 (3.83) | 3.2 (4.15) | 2.4 (3.73) | 2.8 (3.91)
IHS4 Score [Mean (Standard Deviation); unit: score on a scale] — IHS4- International HS Severity Scoring System IHS4 score (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or less signified mild HS, a score of 4-10 signifies moderate HS and a score of 11 or higher signified severe HS.
  score on a scale | 29.6 (29.34) | 33.8 (31.95) | 30.0 (25.02) | 31.2 (28.90)
Subject's Global Assessment of Skin Pain NRS [Mean (Standard Deviation); unit: score on a scale] — NRS- numeric rating scale Subjects recorded the maximum severity pain on a numeric rating scale (NRS) from 0 (no skin pain) to 10 (skin pain as bad as can be imagined) in a daily diary from 1 week before day 1 through the week 44 visit. Population: Baseline characteristic value is not available for all patients.
  score on a scale
    number analyzed (Participants) | 126 | 129 | 127 | 382
    (all) | 5.6 (2.52) | 5.3 (2.54) | 5.2 (2.47) | 5.4 (2.51)
Previous TNF Inhibitor Use [Count of Participants; unit: Participants] — TNF- tumor necrosis factor
  Participants
    Yes | 35 | 38 | 36 | 109
    No | 95 | 96 | 98 | 289
Previously Started (allowed) Concomitant Antibiotic [Count of Participants; unit: Participants]
  Yes | 8 | 9 | 7 | 24
  No | 122 | 125 | 127 | 374

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12.
Description: The percentage of subjects achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12 in the ITT1 population using the NRI-CMH Test. A response was defined as a reduction of at least 50 in abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count compared with baseline.
  The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
  NRI- non-responder imputation; CMH- Cochran-Mantel-Haenszel. Percentage values have been reported as opposed to proportion values to allow for statistical analyses.
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo BID for 12 Weeks
- Avacopan 10 mg: Avacopan 10 mg twice daily (BID) for Period 1+2 of the study
- Avacopan 30 mg: Avacopan 30 mg twice daily (BID) for Period 1+2 of the study
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 130 | 134 | 134
percentage of participants | 30.8 | 22.4 | 35.1
Statistical Analysis 1: Comparison: Placebo vs Avacopan 10 mg; Test type: Other; p = 0.1321, Cochran-Mantel-Haenszel — P-values are obtained from a CMH test stratified by stratification factors Hurley Stage (Stage II vs III), and anti-TNF drug use (Treatment naive vs Previous treatment); % Difference (Avacopan - Placebo) = -8.4, 95% CI 2-sided [-18.7 to 2.4]
Statistical Analysis 2: Comparison: Placebo vs Avacopan 30 mg; Test type: Other; p = 0.4503, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; % Difference (Avacopan - Placebo) = 4.3, 95% CI 2-sided [-6.9 to 15.5]

2. Secondary Outcome: Change From Baseline in Total AN Count at Week 12
Description: The Change from Baseline in total AN (abscess and inflammatory nodule) count at Week 12 using MMRM and OC in the ITT1 population.
  The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
  MMRM - mixed effects model for repeated measures; OC- observed case
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percentage of ANs
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 110 | 110 | 110
percentage of ANs | -3.1 (8.57) | -3.4 (10.58) | -5.1 (8.41)
Statistical Analysis 1: Comparison: Placebo vs Avacopan 10 mg; Test type: Other; p = 0.5784, Mixed model for repeated measures; Least Squares Mean = 0.6, 95% CI 2-sided [-1.7 to 2.9], Standard Error of Mean 1.17
Statistical Analysis 2: Comparison: Placebo vs Avacopan 30 mg; Test type: Other; p = 0.2253, Mixed effects model for repeated measure; Least Squares Mean = -1.4, 95% CI 2-sided [-3.7 to 0.9], Standard Error of Mean 1.17

3. Secondary Outcome: Number of Responders Achieving at Least 30% Reduction and at Least 1 Unit Reduction From Baseline in the Subject's Global Assessment of Skin Pain (NRS30) in Subjects With a Baseline NRS of at Least 3, Evaluated at Week 12
Description: NRS30 = The number of responders achieving at least 30% reduction and at least 1 unit reduction from baseline in the subject's global assessment of skin pain score. Percentage is based on the number of subjects with a baseline pain score of at least 3 in each treatment group.
  Weekly averages of daily pain will be calculated based on subjects' daily diary recording of the worst pain experienced in the previous 24 hours.
  The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
  NRI- non-responder imputation
Time Frame: Baseline to Week 12
Measure: Number; unit: number of responders
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 105 | 104 | 104
number of responders | 26 | 23 | 17

4. Secondary Outcome: Area Under the Curve From Time 0-3hrs (AUC 0-3hrs) of Metabolite M1 Plasma Concentration on Day 1
Description: The Area under the curve from Time 0-3hrs (AUC 0-3hrs) of Metabolite M1 plasma concentration on Day 1 in the PK population.
  PK- pharmacokinetics
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 28 | 29
h*ng/mL | 18.0 (8.23) | 50.3 (34.3)

5. Secondary Outcome: Number of Responders With Baseline Hurley Stage II Who Achieved an AN Count of 0, 1, or 2 at Week 12
Description: The number of responders With Baseline Hurley Stage II Who Achieved an Abscess and Inflammatory Nodule (AN) Count of 0, 1, or 2 at Week 12 using the NRI-CMH Test in the ITT1 population. Hurley Stage II disease is defined as having 1 or more widely separated recurrent abscesses with tract formation and scars.
  The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
Time Frame: Baseline and Week 12
Measure: Number; unit: number of responders
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 85 | 84 | 87
number of responders | 29 | 15 | 20

6. Secondary Outcome: Change of IHS4 Score Relative to Baseline at Week 12.
Description: The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
  IHS4 score (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or less signifies mild HS, a score of 4-10 signifies moderate HS and a score of 11 or higher signifies severe HS.
  IHS4- International HS Severity Scoring System
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 110 | 110 | 110
score on a scale | -6.4 (16.99) | -7.9 (22.14) | -9.8 (15.69)

7. Secondary Outcome: Change From Baseline in Inflammatory Nodule Count at Week 12
Description: A reduction in AN signifies improvement. The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: count of inflammatory nodules
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 110 | 110 | 110
count of inflammatory nodules | -2.4 (7.48) | -2.5 (9.17) | -3.9 (7.06)

8. Secondary Outcome: Change From Baseline in Abscess Count at Week 12
Description: A reduction in abscess count signifies improvement. The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: count of abscesses
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 110 | 110 | 110
count of abscesses | -0.8 (3.68) | -0.8 (3.38) | -1.2 (2.73)

9. Secondary Outcome: Change From Baseline in Draining Fistula Count at Week 12
Description: The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
Time Frame: Baseline and Week 2, Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Draining Fistulae
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 130 | 134 | 134
Draining Fistulae
  Week 2 | -0.3 (2.23) | -0.5 (2.22) | -0.4 (1.79)
  Week 4 | -0.5 (2.17) | -0.8 (2.88) | -0.4 (2.16)
  Week 8 | -0.4 (1.82) | -0.9 (2.93) | -0.6 (2.03)
  Week 12 | -0.6 (2.11) | -0.9 (2.57) | -0.5 (1.87)

10. Secondary Outcome: Change From Baseline to Week 12 in the Modified Sartorius Score to Quantify the Severity Change of HS
Description: Twelve body areas will be evaluated to calculate the Sartorius and modified Sartorius scores: left and right axillae, left and right inframammary areas, intermammary area, left and right buttocks, left and right inguinocrural folds, perianal area, perineal area, and other. The presence of nodules, abscesses, fistulae, scars, and other findings will be recorded. The longest distance between two lesions and whether lesions are separated by normal skin is recorded. A score of 4 indicates the least severe disease, and higher scores indicate increasingly severe disease. There is no upper limit in the score. The ITT1 population was defined as all subjects who were randomized at baseline and received at least 1 dose of investigational product during period 1.
Time Frame: Baseline and Week 2, Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Avacopan 10 mg | Avacopan 30 mg
Number analyzed (Participants) | 130 | 134 | 134
score on a scale
  Week 2 | -3.0 (21.02) | -3.5 (16.68) | -6.3 (17.72)
  Week 4 | -5.7 (23.70) | -7.2 (22.84) | -6.5 (21.37)
  Week 8 | -9.8 (32.60) | -11.5 (23.64) | -10.4 (26.43)
  Week 12 | -11.2 (35.69) | -12.6 (25.98) | -14.4 (29.96)

ADVERSE EVENTS:
Time Frame: All subjects in Period 1 +2 of the study through completion of study an average of 44 weeks
Description: The Safety 1 population was the same as the ITT1 except subjects were assigned to the treatment they received; 1 subject randomized to the placebo group received Avacopan 30 mg during period 1. Thus, this subject is counted in the groups "Avacopan 30 mg Period 1" and "Avacopan 30 mg Period 2" instead of in groups "Placebo Period 1" and "Placebo to Avacopan 30 mg Period 2", respectively
Groups:
- Placebo Period 1: Subjects randomized to placebo during period 1
- Avacopan 10 mg Period 1: Avacopan 10 mg twice daily (BID) for Period 1 of the study
- Avacopan 30 mg Period 1: Avacopan 30 mg twice daily (BID) for Period 1 of the study
- Placebo to Avacopan 10 mg Period 2: Placebo population from Period 1 split into Placebo to Avacopan 10 mg twice daily (BID) for Period 2 of the study
- Placebo to Avacopan 30 mg Period 2: Placebo population from Period 1 split into Placebo to Avacopan 30 mg twice daily (BID) for Period 2 of the study
- Avacopan 10 mg Period 2: Avacopan 10 mg twice daily (BID) for Period 2 of the study
- Avacopan 30 mg Period 2: Avacopan 30 mg twice daily (BID) for Period 2 of the study
Arm/Group | Placebo Period 1 | Avacopan 10 mg Period 1 | Avacopan 30 mg Period 1 | Placebo to Avacopan 10 mg Period 2 | Placebo to Avacopan 30 mg Period 2 | Avacopan 10 mg Period 2 | Avacopan 30 mg Period 2
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/134 | 0/135 | 0/56 | 0/52 | 0/108 | 0/109
Serious Adverse Events (participants affected / at risk) | 3/129 | 3/134 | 1/135 | 0/56 | 1/52 | 4/108 | 2/109
Other Adverse Events (participants affected / at risk) | 22/129 | 18/134 | 15/135 | 7/56 | 8/52 | 21/108 | 20/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Period 1 (N=129) | Avacopan 10 mg Period 1 (N=134) | Avacopan 30 mg Period 1 (N=135) | Placebo to Avacopan 10 mg Period 2 (N=56) | Placebo to Avacopan 30 mg Period 2 (N=52) | Avacopan 10 mg Period 2 (N=108) | Avacopan 30 mg Period 2 (N=109)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculin test false positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Period 1 (N=129) | Avacopan 10 mg Period 1 (N=134) | Avacopan 30 mg Period 1 (N=135) | Placebo to Avacopan 10 mg Period 2 (N=56) | Placebo to Avacopan 30 mg Period 2 (N=52) | Avacopan 10 mg Period 2 (N=108) | Avacopan 30 mg Period 2 (N=109)
Hidradenitis (Skin and subcutaneous tissue disorders) | 17 (35) | 14 (15) | 12 (23) | 5 (6) | 8 (12) | 19 (30) | 19 (31)
Headache (Nervous system disorders) | 4 (10) | 8 (8) | 4 (4) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 5 (6) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03852472/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03852472/SAP_001.pdf